CLINICAL TRIAL: NCT05404516
Title: Prospective Evaluation of Sorafenib Combined With Standard Therapy in Newly Diagnosed Adult Core-binding Factor Acute Myeloid Leukemia: an Open-label , Randomised Controlled, Multicenter Phase II Trial
Brief Title: Combination of Sorafenib With Standard Therapy in Newly Diagnosed Adult CBF AML
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Collaborators: Guangzhou First People's Hospital (Other); Guangzhou Panyu Central Hospital (Other); Institute of Hematology & Blood Diseases Hospital, China (Other); Peking University People's Hospital (Other); Shenzhen Hospital of Southern Medical University (Other); Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Qifa Liu, Professor, Nanfang Hospital, Southern Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Sorafenib-CBF AML-2022
Record Dates: First submitted 2022-05-31; First posted 2022-06-03 (Actual); Last update posted 2022-06-03 (Actual); Status verified 2022-05

CONDITIONS: Core Binding Factor Acute Myeloid Leukemia
Keywords: Core Binding Factor Acute Myeloid Leukemia; Sorafenib; CMR (Complete Molecular Remission)
MeSH Terms: interventions — Sorafenib; Idarubicin; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sorafenib (Experimental): Induction cycle(s):
  IA3+7. Patients will receive sorafenib 400 mg BID on days 8-21.
  Consolidation Cycle 1:
  IA3+3. Patients will receive sorafenib 400 mg BID on days 1-21.
  Consolidation Cycles 2-4:
  MDAC. Patients will receive sorafenib 400 mg BID on days 1-21.
  Maintenance therapy:
  Single agent sorafenib 400 mg BID for one year.
  Interventions: Drug: Sorafenib; Drug: Idarubicin; Drug: Cytarabine
- Standard therapy (Active Comparator): Induction cycle(s):
  IA3+7.
  Consolidation Cycle 1:
  IA3+3.
  Consolidation Cycles 2-4:
  MDAC.
  Interventions: Drug: Idarubicin; Drug: Cytarabine

INTERVENTIONS:
Drug: Sorafenib — Induction cycle(s): 400 mg BID on days 8-21.
  Consolidation cycles 1-4: 400 mg BID on days 1-21.
  Maintenance therapy: 400 mg BID for one year.
  Arms: Sorafenib
Drug: Idarubicin — Induction cycle(s): 12 mg/m2/day on days 1-3.
  Consolidation cycle 1: 8 mg/m2/day administered on days 1-3.
Drug: Cytarabine — Induction cycle(s): 100 mg/m2 by continuous IV infusion for 24 hours on days 1-7.
  Consolidation cycles 1-4: 2 g/m2/12h on days 1-3.

SUMMARY:
Core-binding factor acute myeloid leukemia accounts for 10-15% of AML and is categorized as favorable-risk AML. However, the 5-year CIR was up to 40% in this group of patients. Emerging data show that a high frequency of mutations and/or high expression of KIT in CBF AML. Sorafenib is a multitargeted TKI, thus the purpose of this study is to evaluate the safety and efficacy of sorafenib combined with standard therapy in CBF AML.

DETAILED DESCRIPTION:
Core-binding factor acute myeloid leukemia is characterized by t(8;21) or inv(16) and accounts for 10-15% of AML. Because of the high CR rate of nearly 90% and a 5-year OS of almost 50%, CBF-AML is categorized as favorable-risk AML. However, the 5-year cumulative incidence of relapse (CIR) was up to 40% in this group of patients after high-dose cytarabine consolidation following CR. Therefore, more effective therapeutic approaches are needed.

Emerging data show that a high frequency of mutations and/or high expression of KIT in CBF AML likely result in aberrant tyrosine kinase activity, leukemia cell growth and survival, and treatment resistance. Thus, pharmacologic inhibition of KIT would lead to significant antileukemia activity if combined with an optimized chemotherapy regimen in patients with CBF AML. Recent mechanistic findings also support the potential clinical benefit of KIT inhibition in CBF AML.

Sorafenib is a first-generation type-II multitargeted tyrosine kinase receptor inhibitor (TKI) that suppresses various signaling pathways associated with the development of AML, such as RTK (FLT3, c-KIT), RAS/RAF, vascular endothelial growth factor (VEGF) receptor. The purpose of this study is to evaluate the safety and efficacy of sorafenib combined with standard therapy in CBF AML.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have an unequivocal diagnosis of de novo-CBF AML, prior to start therapy, documented by rearrangement of Core Binding Factor (CBF) genes, namely RUNX1/RUNX1T1 and CBFB/MYH11.
* Age 18 to 65 years old with ECOG performance status 0-2.
* Sign informed consent form, have the ability to comply with study and follow-up procedures.
* Patients must have Total Bilirubin ≤ 1.5 x ULN, and AST or ALT ≤ 2.5 x ULN.
* Patients must have Serum Creatinine ≤ 1.5 x ULN.
* Women of child-bearing potential must have a negative pregnancy test before starting the protocol.

Exclusion Criteria:

* Prior therapy for AML with the following exceptions:

  1. emergency leukapheresis
  2. emergency treatment for hyperleukocytosis with hydroxyurea for ≤ 7 days.
* Central nervous system involvement.
* Presence of any uncontrolled bacterial, viral or fungal infection.
* Known human immunodeficiency virus (HIV) positive.
* An active Hepatitis B virus (HBV) or Hepatitis C virus (HCV) infection. Patients whose disease is controlled under antiviral therapy should not be excluded.
* Presence of other active malignancies.
* QTc > 470 msec (Bazett formula) on screening ECG.
* Presence of significant uncontrolled or active cardiovascular disease, specifically including, but not restricted to:

  1. Myocardial infarction, unstable angina and/or congestive heart failure within 3 months prior to randomization
  2. History of clinically significant (as determined by the treating physician) atrial arrhythmia or any ventricular arrhythmia
  3. Uncontrolled hypertension
  4. Taking medications that are known to be associated with Torsades de Pointes.
* History of hypersensitivity to any drugs or metabolites of similar chemical classes as the study treatment.
* Intolerance to sorafenib, namely persistence of sorafenib-related adverse events despite supportive treatment, persistence or recurrence of adverse events after dose interruption or dose reduction of sorafenib, or both of these.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-08-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
CMR (Complete Molecular Remission) | 1 year
  CMR in BM after 4 cycles of chemotherapies

SECONDARY OUTCOMES:
Overall survival | 3 year
Leukemia-free survival | 3 year
Cumulative incidence of relapse | 3 year
Adverse effects | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Qifa Liu, Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (1):
- Department of Hematology,Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Rucker FG, Agrawal M, Corbacioglu A, Weber D, Kapp-Schwoerer S, Gaidzik VI, Jahn N, Schroeder T, Wattad M, Lubbert M, Koller E, Kindler T, Gotze K, Ringhoffer M, Westermann J, Fiedler W, Horst HA, Greil R, Schroers R, Mayer K, Heinicke T, Krauter J, Schlenk RF, Thol F, Heuser M, Ganser A, Bullinger L, Paschka P, Dohner H, Dohner K. Measurable residual disease monitoring in acute myeloid leukemia with t(8;21)(q22;q22.1): results from the AML Study Group. Blood. 2019 Nov 7;134(19):1608-1618. doi: 10.1182/blood.2019001425. PMID 31554635
- [Background] Paschka P, Schlenk RF, Weber D, Benner A, Bullinger L, Heuser M, Gaidzik VI, Thol F, Agrawal M, Teleanu V, Lubbert M, Fiedler W, Radsak M, Krauter J, Horst HA, Greil R, Mayer K, Kundgen A, Martens U, Heil G, Salih HR, Hertenstein B, Schwanen C, Wulf G, Lange E, Pfreundschuh M, Ringhoffer M, Girschikofsky M, Heinicke T, Kraemer D, Gohring G, Ganser A, Dohner K, Dohner H. Adding dasatinib to intensive treatment in core-binding factor acute myeloid leukemia-results of the AMLSG 11-08 trial. Leukemia. 2018 Jul;32(7):1621-1630. doi: 10.1038/s41375-018-0129-6. Epub 2018 Apr 17. PMID 29720733
- [Background] Rollig C, Serve H, Huttmann A, Noppeney R, Muller-Tidow C, Krug U, Baldus CD, Brandts CH, Kunzmann V, Einsele H, Kramer A, Schafer-Eckart K, Neubauer A, Burchert A, Giagounidis A, Krause SW, Mackensen A, Aulitzky W, Herbst R, Hanel M, Kiani A, Frickhofen N, Kullmer J, Kaiser U, Link H, Geer T, Reichle A, Junghanss C, Repp R, Heits F, Durk H, Hase J, Klut IM, Illmer T, Bornhauser M, Schaich M, Parmentier S, Gorner M, Thiede C, von Bonin M, Schetelig J, Kramer M, Berdel WE, Ehninger G; Study Alliance Leukaemia. Addition of sorafenib versus placebo to standard therapy in patients aged 60 years or younger with newly diagnosed acute myeloid leukaemia (SORAML): a multicentre, phase 2, randomised controlled trial. Lancet Oncol. 2015 Dec;16(16):1691-9. doi: 10.1016/S1470-2045(15)00362-9. Epub 2015 Nov 6. PMID 26549589